CLINICAL TRIAL: NCT01615172
Title: Cannulation of the Artery Axiliaris for Extracorporeal Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Pitzer Stiftung (Unknown)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Cardia vascular research, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AXI-001
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Neurologic Manifestations
MeSH Terms: conditions — Neurologic Manifestations | interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aortic cannulation (Active Comparator): routine placement of aortic cannula
  Interventions: Procedure: cannulation
- axilaris cannulation (Active Comparator): new type of cannulation
  Interventions: Procedure: cannulation

INTERVENTIONS:
Procedure: cannulation — The different types of cannulation (aortic versus axillaris) were compared in the postoperative period for neurological deficits in three time periods.(intraoperative, 5.POD, 3 month POD)
  Other Names: MAQUET 20, 22 and 24 Fr

SUMMARY:
Comparision of two different cannulation techniques on the neurological outcome in cardiac surcical procedures. Study hypothesis: Cannulation of the axilaris artery can reduce neurolocical side effects.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac procedure with ecc Age 40-85 years CABG and/or valve

Exclusion Criteria:

* Stenosis of a.subclavia

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Surrogat endpoint: Number of participants with change from baseline in Neurolocial events at 5th postoperative day (POD) and 3 month after operation | Participants will be followed for the duration of hospital stay (5 POD) and a follow up visit 3 months after discharge
  Neurological events were detected by:NIRO (Near-infrared spectroscopy), EEG (Electrencenphalographie), MRI (Magnet resonance imaging) and test battery (Mini mental status test, HAWIE-R)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zierer, PD.Dr, Principal Investigator — Goethe University
Locations (1):
- Goethe Universität, Frankfurt am Main, Hesse, Germany